CLINICAL TRIAL: NCT00008047
Title: Multicentre Phase II Study Of Concomitant Radio-Chemotherapy Associating Continuous Infusion 5-FU With Hydroxyuree Via Bone Marrow With Or Without Paclitaxel In Treatment Of Inoperable Epidermoid Carcinoma Of Esophagus
Brief Title: Combination Chemotherapy Combined With Radiation Therapy in Treating Patients Who Have Stage II or Stage III Cancer of the Esophagus
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068368; FRE-GERCOR-D99-1; EU-20021
Record Dates: First submitted 2001-01-06; First posted 2003-01-27 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2001-02

CONDITIONS: Esophageal Cancer
Keywords: stage II esophageal cancer; stage III esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Fluorouracil; Hydroxyurea; Paclitaxel; Radiotherapy

INTERVENTIONS:
Drug: fluorouracil
Drug: hydroxyurea
Drug: paclitaxel
Procedure: conventional surgery
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining more than one chemotherapy drug with radiation therapy may kill more tumor cells.

PURPOSE: Randomized phase I/II trial to study the effectiveness of combination chemotherapy with or without paclitaxel combined with radiation therapy in treating patients who have stage II or stage III cancer of the esophagus.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of concurrent radiotherapy with fluorouracil and hydroxyurea with or without paclitaxel in terms of survival without dysphagia in patients with inoperable stage II or III epidermoid carcinoma of the esophagus.
* Compare the overall survival, response rate, toxicity, and quality of life in this patient population treated with these regimens.

OUTLINE: This is a randomized, open label, multicenter study. Patients are stratified according to weight loss (less than 10% vs at least 10%) and inoperability criteria (nonresectable vs due to anatomical terrain). Patients are randomized to one of two treatment arms.

* Arm I: Patients receive fluorouracil IV continuously, oral hydroxyurea, and concurrent radiotherapy daily on days 1-5.
* Arm II: Patients receive fluorouracil, hydroxyurea and radiotherapy as in arm I. Patients also receive paclitaxel IV on day 1.

Treatment continues every 2 weeks for 4 courses in the absence of disease progression or unacceptable toxicity.

Patients with possible resectable disease undergo surgical resection at 4-6 weeks following the last course of chemoradiotherapy. Patients with continued unresectable disease receive 2 additional courses of chemoradiotherapy as above within 8-17 days following the last course of chemoradiotherapy.

Quality of life is assessed at baseline, monthly during therapy, every 2 months for 6 months, every 4 months for 1 year, and then every 6 months thereafter.

Patients are followed every 2 months for 6 months, every 4 months for 1 year, and then every 6 months thereafter.

PROJECTED ACCRUAL: A maximum of 90 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage II (T2 or T3, N0, M0) or III (T3, N1, M0) epidermoid carcinoma of the esophagus
* Inoperable due to initial extension or inoperable with no extension
* No visceral metastases
* No extension to the tracheo-bronchial pathway

  * No tracheo-esophageal fistula
  * No broncho-esophageal fistula
  * No suspected respiratory mucosal involvement on bronchoscopy
* No carcinoma in situ

PATIENT CHARACTERISTICS:

Age:

* 18 to 80

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Platelet count at least 120,000/mm^3
* Hemoglobin at least 10 g/dL
* Neutrophil count at least 1,500/mm^3
* Lymphocyte count at least 1,000/mm^3

Hepatic:

* SGOT and SGPT no greater than 2 times normal
* Albumin at least 3.0 g/dL

Renal:

* Creatinine no greater than 1.4 mg/dL
* Calcium less than 11.2 mg/dL

Pulmonary:

* See Disease Characteristics
* No severe respiratory illness (e.g., severe broncho-pathway obstruction or insufficient respiration)
* No uncontrolled broncho-pulmonary infection

Other:

* No other prior history of malignancy except curatively treated carcinoma in situ of the colon or skin cancer
* No contraindication to fluorouracil
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No psychiatric illness
* HIV negative
* Total protein at least 65% of normal

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior biologic therapy

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* No prior endocrine therapy

Radiotherapy:

* No prior radiotherapy

Surgery:

* See Disease Characteristics

Other:

* No concurrent participation in other study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-08

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Ganem, MD, Study Chair — Centre Jean Bernard
Locations (14):
- France (14):
  - Hopital Saint-Louis, Amiens
  - Clinique Saint Vincent, Besançon
  - Clinique Saint - Jean, Cagne-sur-Mer
  - CHR de Grenoble - La Tronche, Grenoble
  - Hopital Andre Mignot, Le Chesnay
  - CMC Les Ormeaux, Le Havre
  - Centre Jean Bernard, Le Mans
  - Hopital Laennec, Paris
  - Hopital Saint Antoine, Paris
  - Hopital Tenon, Paris
  - Clinique Ste - Marie, Pontoise
  - Polyclinique De Courlancy, Reims
  - C.H. Senlis, Senlis
  - Clinique Fleming, Tours